CLINICAL TRIAL: NCT06972342
Title: Fit & Active Retirement: A Mobile-based, Combined Coach- and Peer-led Physical Function Programme for Young-old Retirees
Brief Title: Fit & Active Retirement: A Physical Function Programme for Young-old Retirees
Acronym: Fit&Active
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Amy S. Ha, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KPF23GWP21
Record Dates: First submitted 2025-01-20; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: balance; muscular strength; retired adults
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- physical functions intervention (Experimental): All participants will take part in base line test, intervention and post-test. The interventions include coach-led co-activity sessions (virtual or in-person), online videos, peer group.
  Interventions: Behavioral: education

INTERVENTIONS:
Behavioral: education — Participants will be intervened after the baseline measurements, including two training classes.

SUMMARY:
Physical inactivity is the fourth leading cause of mortality in the world; as such, the World Health Organization (WHO) recommends that adults engage in at least 150 minutes of moderate-intensity physical activity every week. In addition, the WHO further recommends that older adults (i.e., those 65 years or above) engage in activities that promote functional balance and muscular strength to reduce the risks of falls. This is important because falls are the leading cause of injury-related deaths among older adults. Research has also shown that having good physical function (i.e., activity level, balance, and strength) is associated with better health, well-being, and quality of life. As suggested by results from the Hong Kong Health Behaviour Survey 2018/19, older adults in Hong Kong are generally active, with 85% of the population doing more than 150 minutes of activity on a weekly basis. The survey, however, did not include questions about whether respondents engaged in functional balance training. The above figures suggest that older adults may be unaware of the importance of functional balance and strength training and may not be attaining their optimal levels of physical function. Our proposed study aims to address this issue by delivering an intervention program aimed at increasing retirees' physical activity levels, with emphasis placed on functional balance and muscular strength training. Retirees in Hong Kong are generally healthy, active, and capable of self-learning and self-regulation. Provision of knowledge and support could lead to positive behavior change. Also, as mobile-based messaging (e.g., WhatsApp) has become mainstream, retirees have a good level of competence in using mobile phones as a means of communication. This mode of communication has become increasingly important since face-to-face contact could be impeded by pandemic-led social distancing. Therefore, the proposed project will be delivered primarily through e-platforms. Our previous work has shown that adults' behaviors and attitudes could be enhanced through an internet-based program. Preliminary results of our ongoing retiree-focused program also suggest that older adults are receptive to mobile-based interventions.

DETAILED DESCRIPTION:
A series of educational videos will be produced and placed on the project website to provide participants with knowledge on the importance of having good physical function. Coach-led videos will also be produced for participants to exercise by following on-screen instructions. The exercises included will incorporate activities to improve activity levels, functional balance, and muscular strength. To maximize adherence, a group of participants will first be recruited and trained to serve as "captains" of the program. Each captain will then be assigned to lead a group of participants (5 to 10), ideally recruited through their own social circles, where they will coordinate co-activity sessions (virtual or in-person) by following the provided materials together. Research using a similar peer-led mode has been found to be effective in enhancing behavior and increasing perceived support.

ELIGIBILITY:
Inclusion Criteria:

* healthy, retired and do not have full-time job

Exclusion Criteria:

-

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 300 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Moderate-to-vigorous physical activity | baseline, 2-week before intervention
  measured by ActiGraph GT3X+. The unit of measure is the mean time spent in MVPA per day. Participants will be asked to wear the devices on their waist over a seven-day period, except during water-based activities. Data will be considered valid if participants worn the devices for eight hours on at least two weekdays and one weekend day. Age-appropriate cut-off values will be used for PA intensity classification, i.e., cutpoints by Freedson, Melanson, and Sirard (1998). The mean time participants spent in MVPA during valid days will be used as a measure for MVPA.
Moderate-to-vigorous physical activity | 4 months
  measured by ActiGraph GT3X+. The unit of measure is the mean time spent in MVPA per day. Participants will be asked to wear the devices on their waist over a seven-day period, except during water-based activities. Data will be considered valid if participants worn the devices for eight hours on at least two weekdays and one weekend day. Age-appropriate cut-off values will be used for PA intensity classification, i.e., cutpoints by Freedson, Melanson, and Sirard (1998). The mean time participants spent in MVPA during valid days will be used as a measure for MVPA.
Lower limb strength | baseline, 2-week before intervention
  Use handheld dynamometer to test partipants lower limb strength. Two trials for each leg.
Lower limb strength | 4 months
  Use handheld dynamometer to test partipants lower limb strength. Two trials for each leg.
Upper limb strength | baseline, 2-week before intervention
  Hand grip strength test will also be used as a measure of upper limb strength of participants.
Upper limb strength | 4 months
  Hand grip strength test will also be used as a measure of upper limb strength of participants.
Muscular strength | baseline, 2-week before intervention
  The tests for lower limb strength, reaction time, and standing balance from the Physiological Profile Assessment will also be administered to participants. Hand grip strength test will also be used as a measure of upper limb strength of participants.
Muscular strength | 4 months
  The tests for lower limb strength, reaction time, and standing balance from the Physiological Profile Assessment will also be administered to participants. Hand grip strength test will also be used as a measure of upper limb strength of participants.

SECONDARY OUTCOMES:
The Timed Up and Go test | baseline, 2-week before intervention
  The Timed Up and Go test will be used to assess the level of balance in adults. Participants will be timed as they stand up from a standard armchair, walk 3 meters away, and return. An older adult who takes ≥12 seconds to complete the TUG is at risk for falling
The Timed Up and Go test | 4 months
  The Timed Up and Go test will be used to assess the level of balance in adults. Participants will be timed as they stand up from a standard armchair, walk 3 meters away, and return. An older adult who takes ≥12 seconds to complete the TUG is at risk for falling
The Sit-to-Stand Test | baseline, 2-week before intervention
  The Sit-to-Stand Test, requires participants to repeatedly sit down and stand up as quickly as possible. The time required to complete five repetitions will be used as the score for the test.
The Sit-to-Stand Test | 4 months
  The Sit-to-Stand Test, requires participants to repeatedly sit down and stand up as quickly as possible. The time required to complete five repetitions will be used as the score for the test.
The Four Stage Balance Test | baseline, 2-week before intervention
  The four stage balance test requires participants to stand in a side-by-side-stance, semi-Tandem stance, and a full Tandem stance. The time participants could maintain in a balance position will be scored using a specific scoring rubric. Not being able to hold the tandem stance (task number 3) for 10 seconds is an indication of increased risk of fall.
The four stage balance test | 4 months
  The four stage balance test requires participants to stand in a side-by-side-stance, semi-Tandem stance, and a full Tandem stance. The time participants could maintain in a balance position will be scored using a specific scoring rubric. Not being able to hold the tandem stance (task number 3) for 10 seconds is an indication of increased risk of fall.
Gait pattern | baseline, 2-week before intervention
  Participants' gait pattern will be assessed by GAITRite system walkway. Participants will be asked to walk as usual on a 4.6m long mat twice.
Gait pattern | 4 months
  Participants' gait pattern will be assessed by GAITRite system walkway. Participants will be asked to walk as usual on a 4.6m long mat twice.
Hand reaction time | baseline, 2-week before intervention
  Participants' dominant hand reaction time will be assessed by the reaction timer. Participants will be asked to pay attention to the light on a mouse. Once the light is on, participants should press the button on the mouse as quickly as possible. Ten trials will be conducted.
Hand reaction time | 4 months
  Participants' dominant hand reaction time will be assessed by the reaction timer. Participants will be asked to pay attention to the light on a mouse. Once the light is on, participants should press the button on the mouse as quickly as possible. Ten trials will be conducted.
Life satisfaction | baseline, 2-week before intervention
  Life satisfaction will be measured by WHOQOL-BREF (World Health Organization Quality of Life-BREF) questionnaire. Twenty-six items will be rated on a 5-point Likert scale, ranging from 1 (not at all) to 5 (completely). All items will be added up including Item 3 will be reverse-coded first. Higher total scores indicate a higher quality of life.
Life satisfaction | 4 months
  Life satisfaction will be measured by WHOQOL-BREF (World Health Organization Quality of Life-BREF) questionnaire. Twenty-six items will be rated on a 5-point Likert scale, ranging from 1 (not at all) to 5 (completely). All items will be added up including Item 3 will be reverse-coded first. Higher total scores indicate a higher quality of life.
Social support for exercise | baseline, 2-week before intervention
  Social support for exercise is assessed by Social Support and Exercise Survey. Higher scores indicate higher support from family and friends on exercise.
Social support for exercise | 4 months
  Social support for exercise is assessed by Social Support and Exercise Survey. Higher scores indicate higher support from family and friends on exercise.
eHealth Literacy | baseline, 2-week before intervention
  eHealth Literacy is assessed by eHealth Literacy Scale (eHEALS）. Higher scores of eight items indicate better eHealth Literacy.
eHealth Literacy | 4 months
  eHealth Literacy is assessed by eHealth Literacy Scale (eHEALS）. Higher scores of eight items indicate better eHealth Literacy.
Perceived falling risk | baseline, 2-week before intervention
  Participants are asked to report how much they are concerned about falling when engaging in seven daily activities, e.g.take on/off clothes, taking bath/shower. Higher total scores on seven items indicate higher perceived falling risk.
Perceived falling risk | 4 months
  Participants are asked to report how much they are concerned about falling when engaging in seven daily activities, e.g.take on/off clothes, taking bath/shower. Higher total scores on seven items indicate higher perceived falling risk.
Self-report physical activity frequency | baseline, 2-week before intervention
  Participants are asked to answer two items about how frequent they engage in PA to enhance muscular strength and functional balance.
Self-report physical activity frequency | 4 months
  Participants are asked to answer two items about how frequent they engage in PA to enhance muscular strength and functional balance.
Sports motivation | baseline, 2-week before intervention
  Participants' sports motivation will be measured by 24 items on a five-point scale (0- completely not suitable for me, 4-completely suitable for me), such as I think doing exercise is a joyful thing.
Sports motivation | 4 months
  Participants' sports motivation will be measured by 24 items on a five-point scale (0- completely not suitable for me, 4-completely suitable for me), such as I think doing exercise is a joyful thing.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No